CLINICAL TRIAL: NCT04634331
Title: Dual-task Augmented Reality Treatment for Parkinson's Disease (DART)
Brief Title: Dual-task Augmented Reality Treatment for Parkinson's Disease
Acronym: DART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Jay Alberts, Staff, Department of Biomedical Engineering, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-207
Record Dates: First submitted 2020-11-09; First posted 2020-11-18 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; dual task; postural instability; gait dysfunction
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: 50 individuals with Parkinson's disease will be randomized to either 1) traditional multi-modal training, or 2) augmented reality multi-modal training.
Who Masked: Investigator
Masking Description: The investigator performing the assessments will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Multi-Modal Training (Active Comparator): A physical therapist will provide 1:1 multi-modal training. Multi-modal training is the simultaneous performance of a motor and a cognitive task (i.e. marching while answering math questions)
  Interventions: Behavioral: Traditional Multi-Modal Training
- Augmented Reality Multi-Modal Training (Experimental): Multi-modal training will be administered via the Microsoft HoloLens 2 augmented reality head set. Augmented reality allows user to see the real world, and inserts holograms into the environment. For example, the user could see boxes on the ground that they need to step around when walking. The boxes are not real, but rather a hologram that only the user can see. The augmented reality device will instruct the participant on the motor and cognitive task that should be performed simultaneously in a similar manner to the physical therapist in the traditional multi-modal training group. The intervention will be overseen by a physical therapist.
  Interventions: Behavioral: Augmented Reality Multi-Modal Training

INTERVENTIONS:
Behavioral: Augmented Reality Multi-Modal Training — Training administered via an augmented reality headset.
  Arms: Augmented Reality Multi-Modal Training
Behavioral: Traditional Multi-Modal Training — Training administered via a 1:1 physical therapy session
  Arms: Traditional Multi-Modal Training

SUMMARY:
Activities of daily living (ADL) frequently involve the simultaneous performance of two or more tasks, such as crossing the street while holding a conversation, commonly referred to as dual tasking. The simultaneous performance of a motor and a cognitive task increases postural instability, gait dysfunction, and may increase fall rates in Parkinson's disease (PD). The goal of this project is to evaluate the effectiveness of utilizing a digital therapeutic, Dual-task Augmented Reality Treatment (DART) protocol, for the treatment of postural instability and gait dysfunction (PIGD) in individuals with PD. A randomized controlled trial will be conducted at the Main Campus of the Cleveland Clinic (Cleveland, OH). A total of 50 individuals with Parkinson's disease will be randomized into 1) a traditional multi-modal training group, or 2) multi-modal training administered via an augmented reality headset. Multi-modal therapy is where the participant practices performing two things at once (i.e. marching while answering math questions). Augmented reality is a type of head-worn technology that allows the individual to see the real world and places holograms in the space. Both groups will exercise 2x/week for a total of 8 weeks. Assessments involving walking, balancing, and turning will be completed to assess the efficacy of the treatment.

DETAILED DESCRIPTION:
Individuals with Parkinson's disease who qualify for the study will come to the Cleveland Clinic for an informed consent visit. At the informed consent visit, the participant will receive an activity monitor and a fall diary. Following a 4-week period where activity and falls are monitored, the participant will come to the Cleveland Clinic for a comprehensive physical and cognitive assessment primarily using a virtual reality treadmill system. During that baseline assessment, the individual will be randomized to either 1) traditional multi-modal training, or 2) augmented reality multi-modal training. Regardless of group allocation, the participant will complete a total of 16 treatment sessions (2x/week for 8 weeks). The traditional multi-modal treatment will be administered 1:1 by a physical therapist. The augmented reality multi-modal training will be overseen by a physical therapist and administered via the Microsoft HoloLens 2 augmented reality device. Follow-up assessments will be conducted at the end of the 16 treatment sessions and 8 weeks after the treatment sessions have ceased. Falls and activity data will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult with a diagnosis of idiopathic PD
2. Self-reported gait or balance deficits
3. Hoehn and Yahr stage I-III
4. Ability to ambulate >10 minutes continuously

Exclusion Criteria:

1. Diagnosis of dementia or any neurocognitive impairment that compromises the ability to provide informed consent
2. >2 errors on the Short Portable Mental Status Questionnaire
3. Implanted deep brain stimulation electrodes
4. Musculoskeletal or cardiopulmonary issue that limits one's ability to engage in exercise
5. Neurological disease other than Parkinson's disease that impacts motor or cognitive function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Alberts, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alberts JL, Kaya RD, Penko AL, Streicher M, Zimmerman EM, Davidson S, Walter BL, Rosenfeldt AB. A Randomized Clinical Trial to Evaluate a Digital Therapeutic to Enhance Gait Function in Individuals With Parkinson's Disease. Neurorehabil Neural Repair. 2023 Sep;37(9):603-616. doi: 10.1177/15459683231184190. Epub 2023 Jul 19. PMID 37465959

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Traditional Multi-Modal Training | Augmented Reality Multi-Modal Training
Started | 24 | 27
Completed | 22 | 25
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Multi-Modal Training | Augmented Reality Multi-Modal Training | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 18 | 22 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (6.1) | 69.9 (6.2) | 69.2 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 16 | 22 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black | 2 | 3 | 5
  White | 21 | 23 | 44
Region of Enrollment [Number; unit: participants]
  United States | 24 | 27 | 51

OUTCOME MEASURES:

1. Primary Outcome: Gait Velocity
Description: Walking speed (m/s) on a self-paced treadmill during single and dual task conditions
Time Frame: From baseline assessment to the end of the 8-week training session
Measure: Mean (Standard Error); unit: meters/second
Arm/Group | Traditional Multi-Modal Training | Augmented Reality Multi-Modal Training
Number analyzed (Participants) | 22 | 25
meters/second
  Baseline Single-task Walk Speed | 1.20 (0.19) | 1.22 (0.20)
  Baseline Serial 7 Dual-Task Walk Speed | 1.03 (0.24) | 1.07 (0.29)
  Baseline Digit Recall Dual-Task Walk Speed | 1.05 (0.18) | 1.09 (0.23)
  Baseline Controlled Oral Word Association Dual-Task Walk Speed | 1.09 (0.19) | 1.11 (0.24)
  Baseline Stroop Dual-Task Walk Speed | 1.11 (0.23) | 1.19 (0.25)
  Baseline 1-Back Dual-Task Walk Speed | 1.07 (0.27) | 1.11 (0.27)
  Baseline 2-Back Dual-Task Walk Speed | 1.08 (0.27) | 1.09 (0.29)
  End of Treatment Single-task Walk | 1.27 (0.19) | 1.33 (0.25)
  End of Treatment Serial 7 Dual-Task Walk Speed | 1.12 (0.23) | 1.22 (0.31)
  End of Treatment Digit Recall Dual-Task Walk Speed | 1.14 (0.22) | 1.22 (0.29)
  End of Treatment Controlled Oral Word Association Dual-Task Walk Speed | 1.17 (0.21) | 1.22 (0.29)
  End of Treatment Stroop Dual-Task Walk Speed | 1.19 (0.25) | 1.27 (0.29)
  End of Treatment 1-Back Dual-Task Walk Speed | 1.18 (0.26) | 1.25 (0.30)
  End of Treatment 2-Back Dual-Task Walk Speed | 1.17 (0.29) | 1.22 (0.33)

2. Primary Outcome: MDS-UPDRS III Score
Description: Global score of motor function in Parkinson's disease using the Movement Disorders Society-Unified Parkinson's Disease Rating Scale subscale III (MDS-UPDRS III). Eighteen items scored on a 0-4 scale resulting in a score ranging from 0-72. A higher score (larger number) indicates more motor symptoms.
Time Frame: From baseline assessment to the end of the 8-week training session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Multi-Modal Training | Augmented Reality Multi-Modal Training
Number analyzed (Participants) | 22 | 25
score on a scale
  Baseline MDS-UPDRS III Score | 34.1 (13.1) | 37.6 (12.3)
  End of Treatment MDS-UPDRS III Score | 34.9 (11.4) | 36.6 (12.8)

3. Primary Outcome: Fall Frequency
Description: number of falls in the previous 30 day period
Time Frame: From baseline assessment to the end of the 8-week training session
Measure: Mean (Standard Deviation); unit: number of falls
Arm/Group | Traditional Multi-Modal Training | Augmented Reality Multi-Modal Training
Number analyzed (Participants) | 22 | 25
number of falls
  Baseline Number of falls | 0.5 (1.22) | 0.68 (1.14)
  End of Treatment Number of Falls | 0.64 (1.59) | 0.52 (0.71)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 5 month study enrollment for each participant.
Arm/Group | Traditional Multi-Modal Training | Augmented Reality Multi-Modal Training
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/27
Other Adverse Events (participants affected / at risk) | 0/24 | 1/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traditional Multi-Modal Training (N=24) | Augmented Reality Multi-Modal Training (N=27)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Participant fell during training session.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traditional Multi-Modal Training (N=24) | Augmented Reality Multi-Modal Training (N=27)
Fall (Injury, poisoning and procedural complications) | NA | 1 (1) — Participant fell during training session.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT04634331/Prot_SAP_000.pdf